CLINICAL TRIAL: NCT07192367
Title: Comparison of the Effectiveness Level of Virtual Reality Exposure Therapy With Sertraline Treatment in Social Anxiety Disorder
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emine Kanmaz (Other)
Collaborators: Kocaeli University (Other)
Responsible Party: Sponsor-Investigator, Emine Kanmaz, Kocaeli University, Department of Child and Adolescent Psychiatry, Kocaeli University
Organization: Kocaeli University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGMBT24; BAP-2024 (Other Grant/Funding Number: Kocaeli University Scientific Research Projects Coordination Unit (BAP)); KAEK/06.bI.08 (Other: Kocaeli University Clinical Research Ethics Committee); 580850 (Other: Kocaeli University Rectorate (Document No: E-89460677-730.99-580850)); 24-AKD-86 (Other: Turkish Medicines and Medical Devices Agency (TITCK))
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Social Anxiety Disorder
Keywords: Social Phobia; Virtual Reality Exposure Therapy; Sertraline; Adolescents; Anxiety Disorders
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders | interventions — Virtual Reality Exposure Therapy; Sertraline; Antidepressive Agents

STUDY DESIGN:
Intervention Model Description: "Participants are assigned to one of two parallel groups: one group receives Virtual Reality Exposure Therapy, and the other group receives Sertraline treatment. The interventions are administered concurrently, without crossover between groups."
Masking Description: This is an open-label study. Neither participants, care providers, investigators, nor outcome assessors are blinded to the intervention assignments. The nature of the interventions (VR exposure therapy vs. sertraline treatment) makes blinding infeasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtual Reality Exposure Therapy (Experimental): RESEARCH ARM: This will be a group of volunteer patients who are being followed up with SAB in our outpatient clinic but who do not accept medication treatment and who will be informed about Virtual Reality Exposure Therapy (VRIT) through a poster presentation.
  Interventions: Behavioral: Virtual Reality Exposure Therapy
- Sertraline (Active Comparator): CONTROL ARM: This will consist of patients who have newly applied to our outpatient clinic and have been diagnosed with Social Anxiety Disorder (SAD), who are the first treatment option in our routine outpatient clinic follow-up, who are deemed appropriate to begin sertraline treatment, and who accept medication treatment.
  Interventions: Drug: Sertraline (Oral Antidepressant)

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy — Participants receive structured Virtual Reality Exposure Therapy sessions using a VR headset. The intervention provides simulated social situations (e.g., public speaking, group interactions) to gradually expose participants to anxiety-provoking scenarios. The sessions are guided and standardized to target symptoms of social anxiety disorder.
  Other Names: VR Therapy; VR Exposure
  Arms: Virtual Reality Exposure Therapy
Drug: Sertraline (Oral Antidepressant) — Participants receive pharmacological treatment with Sertraline, a selective serotonin reuptake inhibitor (SSRI) commonly prescribed for social anxiety disorder. Dosage and administration will follow clinical guidelines and physician judgment.
  Other Names: SSRI; Zoloft
  Arms: Sertraline

SUMMARY:
This study compares two treatment approaches for adolescents and young adults with social anxiety. One group will participate in therapy sessions using a virtual reality headset, while the other group will receive sertraline, a commonly used medication for social anxiety. The goal is to see which treatment is more effective in reducing anxiety symptoms and improving daily functioning. The study will also look at how acceptable and safe these treatments are. A total of 56 participants will be enrolled at Kocaeli University, Department of Child and Adolescent Psychiatry.

DETAILED DESCRIPTION:
Social anxiety disorder (SAD) is a common psychiatric condition that often begins in adolescence and causes significant impairment in academic, social, and occupational functioning. Although selective serotonin reuptake inhibitors (SSRIs) such as sertraline have demonstrated efficacy, many families and patients hesitate to use pharmacological treatments due to concerns about side effects and personal preferences. Virtual reality (VR)-based exposure therapy has emerged as a promising intervention by providing controlled and immersive environments where social situations can be simulated safely.

This study is designed to evaluate the effectiveness of VR exposure therapy compared with sertraline in adolescents and young adults diagnosed with SAD. Participants (N = 56) will be allocated to either VR therapy or sertraline treatment depending on treatment preference. The primary outcome will be reduction in social anxiety symptoms assessed with standardized clinical scales. Secondary outcomes will include functional improvements, treatment acceptability, and safety assessments.

The trial is conducted at Kocaeli University, Department of Child and Adolescent Psychiatry, and aims to provide evidence regarding whether VR exposure therapy can serve as an effective and acceptable alternative to pharmacological treatment in this population.

ELIGIBILITY:
Inclusion Criteria:

* RESEARCH ARM:

  1. Applied to Kocaeli University Child and Adolescent Psychiatry Outpatient Clinic
  2. Have normal intelligence based on clinical observation
  3. Be between 12 and 17 years of age
  4. Have a diagnosis of SAD
  5. Have refused medication recommended for SAD
  6. For SAD; are not currently receiving medical treatment
  7. Have received written consent to participate in the study from them and/or their first-degree relatives authorized to make decisions about them
  8. Have volunteered to participate in the study through an invitation poster presentation

CONTROL ARM:

1 Applied to Kocaeli University Child and Adolescent Psychiatry Outpatient Clinic 2. Have normal intelligence based on clinical observation 3. Be between 12 and 17 years of age 4. Have a diagnosis of SAD 5. Have refused medication recommended for SAD 6. For SAD; are not currently receiving medical treatment 7. Have obtained written informed consent to participate in the study from them and/or their first-degree relatives authorized to make decisions about them 8. Have volunteered to participate in the study through an invitation poster presentation

CONTROL ARM:

1 Applied to Kocaeli University Child and Adolescent Psychiatry Outpatient Clinic 2. Have normal intelligence based on clinical observation 3. Be between 12 and 17 years of age 4. Have a diagnosis of SAD 5. For SAD; Not currently receiving medical treatment 6. Volunteer 7. Written consent for participation in the study must be obtained from the patient and/or their first-degree relative authorized to make decisions about them.

8. Accept sertraline treatment, routinely used in outpatient clinic follow-ups for SAD, and volunteer for the study.

Exclusion Criteria:

RESEARCH ARM:

1. Substance use disorder
2. Schizophrenia and bipolar disorder
3. Autism spectrum disorder
4. Cognitive disability
5. Neurological disorder
6. Balance disorder
7. Patients who have received SSRI treatment for SAD in the last 6 months

CONTROL ARM:

1. Substance use disorder
2. Schizophrenia and bipolar disorder
3. Autism spectrum disorder
4. Cognitive disability
5. Patients who have received SSRI treatment for SAD within the last 6 months -

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Social Anxiety Symptoms (Liebowitz Social Anxiety Scale, LSAS) | Baseline (Week 0), Week 6, and Week 12
  Change from baseline in social anxiety symptoms measured by the Liebowitz Social Anxiety Scale (LSAS). The LSAS evaluates fear and avoidance across 24 items covering social interaction and performance situations, providing total and subscale scores.

SECONDARY OUTCOMES:
Change in Social Phobia Symptoms (Çapa Social Phobia Scale for Children and Adolescents, ÇESFÖ) | Baseline (Week 0), Week 6, and Week 12
  Change from baseline in social phobia symptoms measured by the Çapa Social Phobia Scale for Children and Adolescents (ÇESFÖ), a 25-item self-report Likert-type scale developed for ages 9-17. Higher scores indicate greater severity of social phobia symptoms.
Change in Anxiety Symptoms (Screen for Child Anxiety Related Emotional Disorders, SCARED) | Baseline (Week 0), Week 6, and Week 12
  Change from baseline in anxiety symptoms measured by the Screen for Child Anxiety Related Emotional Disorders (SCARED), including child- and parent-report forms (41 items total, yielding total and subscale scores).

CONTACTS AND LOCATIONS:
Overall Officials: Nursu Çakın Memik, MD, Prof., Principal Investigator — Kocaeli University, Department of Child and Adolescent Psychiatry; Emine Kayış, MD, Study Director — Kocaeli University, Department of Child and Adolescent Psychiatry
Locations (1):
- Kocaeli University Hospital - Department of Child and Adolescent Psychiatry, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because this study is a single-center academic thesis project, and the data contains sensitive personal health information of minors. Data confidentiality and privacy regulations prevent sharing with external researchers.